CLINICAL TRIAL: NCT00940511
Title: Effects of Coordinated Care for Disabled Medicaid Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDRC (Other)
Collaborators: Center for Health Care Strategies (Other); Robert Wood Johnson Foundation (Other); Colorado Department of Health Care Policy and Financing (Unknown); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Charles Michalopoulos, Chief Economist, MDRC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MDRC-CO-02
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Conditions Faced by Medicaid Recipients With Disabilities
Keywords: All conditions faced by disabled Medicaid recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coordinated care (Experimental): Individuals will be passively enrolled in Medicaid managed care. Those who do not opt out of managed care will be provided with care coordination.
  Interventions: Behavioral: Coordinated care
- Usual care (No Intervention): The usual care group will remain in fee-for-service Medicaid and receive services normally available through that system.

INTERVENTIONS:
Behavioral: Coordinated care
  Arms: Coordinated care

SUMMARY:
The purpose of this study is to improve the quality of care for individuals with multiple chronic conditions, health care systems have begun turning to coordinated care. Although coordinated care can refer to many different things, it usually includes activities such as assessing patients' needs, referring them to the right doctors, helping them make and keep appointments, and helping them comply with medical or dietary recommendations. To understand the effects of coordinated care for high-needs Medicaid recipients, MDRC is conducting a randomized trial of a pilot coordinated care program run by Kaiser Permanente for blind and disabled Medicaid recipients in the Denver area.

ELIGIBILITY:
Inclusion Criteria:

* Disabled, in fee-for-service Medicaid

Exclusion Criteria:

* Under age 18, over age 64

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2618 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Health care use through Medicaid | Two years

SECONDARY OUTCOMES:
Primary and preventive care | Six months, two years
Emergency department use | Six months, two years
Hospital admissions | Six months, two years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Michalopoulos, Ph.D., Principal Investigator — MDRC
Locations (1):
- Kaiser Permanente, Jefferson County, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michalopoulos C, Manno MS, Warren A, Somers J. Managing Health Care for Medicaid Recipients with Disabilities: Final Report on the Kaiser Permanente Colorado Coordinated Care Pilot Program. New York: MDRC
- [Result] Kim SE, Michalopoulos C, Kwong RM, Warren A, Manno MS. Telephone care management's effectiveness in coordinating care for Medicaid beneficiaries in managed care: a randomized controlled study. Health Serv Res. 2013 Oct;48(5):1730-49. doi: 10.1111/1475-6773.12060. Epub 2013 Apr 5. PMID 23557249
- See also: Published reports — http://www.mdrc.org/project/coordinated-care-high-cost-medicaid-recipients-disabilities#related_content